CLINICAL TRIAL: NCT05483543
Title: A Prospective, Phase II, Single-arm Study Evaluating the Efficacy and Safety of Pamiparib in Consolidation Therapy for Limited-stage Small Cell Lung Cancer That Has Not Progressed After Concurrent Chemoradiotherapy
Brief Title: Pamiparib for Consolidation Treatment of Unprogressed LS-SCLC After Concurrent Chemoradiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Fudan University, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSSCLCPARPI-01
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Limited Stage Small Cell Lung Cancer
MeSH Terms: interventions — pamiparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pamiparib monoagent (Experimental): Drug: Pamiparib 40mg bid orally
  Interventions: Drug: Pamiparib

INTERVENTIONS:
Drug: Pamiparib — Patients will receive Pamiparib 40 mg bid every 3 weeks after cCRT up to 1 year or disease progression according to RECIST v1.1 occur.
  Other Names: BGB-290

SUMMARY:
This study is a prospective, single-arm, phase II clinical trial, with 1-year PFS as the endpoint, to evaluate the efficacy and associated toxicity of Pamiparib as single-agent consolidation treatment in patients with limited-stage small cell lung cancer(LS-SCLC) patients who have not progressed following platinum-based concurrent chemoradiotherapy(cCRT) .

ELIGIBILITY:
Inclusion Criteria:

* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry, had good compliance and cooperated with the follow-up.
* Age at least 18 years
* Pathologically (histologically or cytologically) proven diagnosis of limited stage small cell lung cancer (Stage Tx, T1-T4, N0-3, M0, American Joint Committee on Cancer [AJCC] staging, 8th edition [Ed.]), within 60 days prior to registration
* Patients must have had measurable disease (per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1) prior to the required cycle of cCRT
* Patients must be free of disease progression and not be able to receive other antitumor therapy within 6 weeks of completion of cCRT
* Patients must submit archived or freshly biopsied tumor tissue (formalin-fixed, paraffin-embedded tissue block or approximately 15 unstained sections [must have >8 sections]) along with the relevant pathology report.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 30 days prior to registration
* Patient life expectancy must be >12 weeks

Exclusion Criteria:

* Mixed SCLC or NSCLC confirmed by histology
* Previous tumor resection for LS-SCLC
* Any patient treatable by surgery or stereotactic body radiation therapy/stereotactic ablative radiation therapy should be excluded
* Expected to receive any other form of anti-tumor therapy during the study period
* Previous treatment with PARP inhibitor drugs
* Any active malignancy within 2 years prior to enrollment, excluding the specific cancers being studied in this study and locally recurrent cancers that have been cured (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, cervical cancer carcinoma in situ or carcinoma in situ of the breast)
* Women who are pregnant, breastfeeding, or planning to become pregnant during the study
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year Progression Free Survival Rate | One year after the start of intervention
  One-year PFS rate was define as the percentage of patients who did not experience disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death due to any cause within 1 year from the date cCRT treatment ended.

SECONDARY OUTCOMES:
Progression Free Survival | Two years
  Progression-free survival according to RECIST v1.1 from date of cCRT treatment ended until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months. For patients whose disease did not progress, PFS was evaluated by censoring patients at their most recent imaging.
Overall Survival | Two years
  Overall survival from date of cCRT treatment ended until the date of end of treatment visit or date of death from any cause, whichever came first, assessed up to 24 months. Participants still alive at the time of data analysis will be censored at the date of last follow-up.
AEs/SAEs | Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first
  The level of AEs defined by NCI-CTCAE v5.0. Safety assessments will be assessed and documented after initiation of study drug, regardless of relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Mao J, Ni J, Chu L, Chu X, Xu D, Yang X, Zhu Z. Pamiparib as consolidation treatment after concurrent chemoradiotherapy of limited-stage small cell lung cancer: a single-arm, open-label phase 2 trial. Radiat Oncol. 2024 Apr 12;19(1):47. doi: 10.1186/s13014-024-02437-2. PMID 38610031